CLINICAL TRIAL: NCT00355602
Title: Use of Antibiotics to Eradicate Bacterial Pathogens Colonising the Colonic Mucosa in Ulcerative Colitis Patients
Brief Title: Antibiotics for the Treatment of Ulcerative Colitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: Tenovus Scotland (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tenovus 134/03
Record Dates: First submitted 2006-07-21; First posted 2006-07-24 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Colitis, Ulcerative
Keywords: Antibiotics; Controlled Clinical Trial
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Cefuroxime; Ciprofloxacin; Clarithromycin; Trimethoprim, Sulfamethoxazole Drug Combination; Amoxicillin-Potassium Clavulanate Combination; Metronidazole; Neomycin; Rifaximin; Vancomycin; Doxycycline

INTERVENTIONS:
Drug: Cefuroxime
Drug: Ciprofloxacin
Drug: Clarithromycin
Drug: Cotrimoxazole
Drug: Coamoxiclav
Drug: metronidazole
Drug: neomycin
Drug: rifaximin
Drug: Vancomycin
Drug: Doxycycline

SUMMARY:
Ulcerative colitis (UC) is an acute and chronic inflammatory bowel disease, whose cause is unknown. However, it is widely accepted that bacteria living in the large bowel are essential for the development of the disease. Intuitively, therefore, a logical approach to treatment would be to use antibiotics. However, antimicrobial chemotherapy has been unsuccessful in managing acute colitis, and has had only limited benefit in long-term treatment. The failure of antibiotics in UC arises from the fact that no-one has tried to identify which bacteria are involved in causing disease, and equally importantly, nobody has targeted appropriate antibiotics to knock out the specific bacteria in question, in a systematic way. Despite this, increasing evidence implicates bacteria living on the lining of the bowel being involved in UC. Our aim, therefore is to identify bacteria colonizing the mucosal surface in the lower large intestine and to determine the antibiotic sensitivities of those the investigators believe to be particularly involved in the disease, such as enterococcit, peptostreptococci and enterobacteria. Because the investigators have already studied resistance to antimicrobial in many mucosal isolate, the investigators plan ot focus on using a combination of two antibiotics in this work. A controlled trial will test the benefit of using these antibiotics over a period of one month and then the patients will be followed up over a six month period. The investigators will be looking for significant long-term improvements, and a reduction in drug use following antibiotic therapy.

DETAILED DESCRIPTION:
It is now widely acknowledged, as a result of experimental studies over the last 30 years, that the mucosal flora of the large bowel are essential to the pathogenesis of ulcerative colitis. Whilst treatment with antibiotics, therefore, might seem a logical approach, a number of clinical trials have proved disappointing. This is because the principal bacteria involved in the inflammatory process have not been identified and their sensitivities to the antibacterials determined. Moreover, we are only now beginning to understand the physiology of biofilm populations on mucosal surfaces, one property of which is antibiotic resistance. Our own studies have show a distinctive bacterial population of the mucosa with UC patients with reduced numbers of protective bifidobacteria and increased enterobacteria which we have linked to disease activity. Antibiotic resistance to commonly used gut antibiotics is widespread in these bacteria.

Our study, therefore, will commence with multiple biopsies of the distal large bowel mucosa being taken in patients with active UC and detailed microbiological characterization of the flora using viable counting, chemotaxonomy and molecular approaches. Antibiotic sensitivities of the likely pathogens will be determined and dissemination of antibiotic resistance genes in the mucosal microbiota followed using real time PCR. Markers of mucosal immune response including proinflammatory cytokines and human betea defensins will also be measured. Two weeks after initial biopsies, the patient will return to pur research IBD clinic where the appropriate combination of antibiotics will be prescribed and these will be taken for one month. A further assessment will occur at the end of this period including mucosal biopsies. endpoints will include clinical activity index, bowel habit diaries, sigmoidoscopy score, mucosal immune markers and routine haematology and biochemical indices. Because of the long term effect of antibiotics on the gut mucosa, which can last for many months, the study cannot be randomised and therefore, the run in period will be taken as a control period and the four weeks on the antibiotic will follow in all patients. The prime endpoint will be sigmoidoscopy score and the subjects will be followed up for a further six months after the study to look for long term benefits.

ELIGIBILITY:
Inclusion Criteria:

* Active ulcerative colitis, CAI greater than or equal to 4

Exclusion Criteria:

* Antibiotics in the last 3 months
* Probiotics
* Alteration to medications in last 3 months

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
sigmoidoscopy score 0,1 and 7 months

SECONDARY OUTCOMES:
mucosal immune markers: human beta defensins, proinflammatory cytokines
haemtaology indices
biochemical indices
clinical activity index
bowel habit diary
all at 0, 1 and 7 months

CONTACTS AND LOCATIONS:
Overall Officials: George T Macfarlane, BSCc, PHD, Principal Investigator — University of Dundee; John H Cummings, MBChB MSc MA, Principal Investigator — University of Dundee; Sandra Macfarlane, BSc, PhD, Principal Investigator — University of Dundee
Locations (1):
- Ninewells Hospital and Medical School, Dundee, Angus, United Kingdom

REFERENCES:
- [Background] Montgomery SM, Morris DL, Thompson NP, Subhani J, Pounder RE, Wakefield AJ. Prevalence of inflammatory bowel disease in British 26 year olds: national longitudinal birth cohort. BMJ. 1998 Apr 4;316(7137):1058-9. doi: 10.1136/bmj.316.7137.1058. No abstract available. PMID 9552907
- [Background] Mayberry JF, Ballantyne KC, Hardcastle JD, Mangham C, Pye G. Epidemiological study of asymptomatic inflammatory bowel disease: the identification of cases during a screening programme for colorectal cancer. Gut. 1989 Apr;30(4):481-3. doi: 10.1136/gut.30.4.481. PMID 2785474
- [Background] Loftus EV Jr, Silverstein MD, Sandborn WJ, Tremaine WJ, Harmsen WS, Zinsmeister AR. Ulcerative colitis in Olmsted County, Minnesota, 1940-1993: incidence, prevalence, and survival. Gut. 2000 Mar;46(3):336-43. doi: 10.1136/gut.46.3.336. PMID 10673294
- [Background] Cummings JH, Macfarlane GT, Macfarlane S. Intestinal bacteria and ulcerative colitis. Curr Issues Intest Microbiol. 2003 Mar;4(1):9-20. PMID 12691258
- [Background] Onderdonk AB, Bartlett JG. Bacteriological studies of experimental ulcerative colitis. Am J Clin Nutr. 1979 Jan;32(1):258-65. doi: 10.1093/ajcn/32.1.258. No abstract available. PMID 760501
- [Background] Macfarlane S, Furrie E, Cummings JH, Macfarlane GT. Chemotaxonomic analysis of bacterial populations colonizing the rectal mucosa in patients with ulcerative colitis. Clin Infect Dis. 2004 Jun 15;38(12):1690-9. doi: 10.1086/420823. Epub 2004 May 25. PMID 15227614
- [Background] Furrie E, Macfarlane S, Kennedy A, Cummings JH, Walsh SV, O'neil DA, Macfarlane GT. Synbiotic therapy (Bifidobacterium longum/Synergy 1) initiates resolution of inflammation in patients with active ulcerative colitis: a randomised controlled pilot trial. Gut. 2005 Feb;54(2):242-9. doi: 10.1136/gut.2004.044834. PMID 15647189